CLINICAL TRIAL: NCT02645123
Title: Gait Analysis of Chronic Low Back Pain Patients Before and After the Application of Spinal Mobilization
Brief Title: Gait in Low Back Pain Patients After Spinal Mobilization
Acronym: SpinMob
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ioannina (Other)
Responsible Party: Principal Investigator, Georgios Krekoukias, Physiotherapist MSc PhD MMACP, University of Ioannina
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 721α/11-10-2011
Record Dates: First submitted 2015-12-23; First posted 2016-01-01 (Estimated); Results first posted 2017-06-08 (Actual); Last update posted 2017-06-08 (Actual); Status verified 2017-05

CONDITIONS: Chronic Low Back Pain
Keywords: spinal mobilization; manual therapy; gait analysis; low back pain; chronic
MeSH Terms: conditions — Low Back Pain; Bronchiolitis Obliterans Syndrome | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Spinal mobilization (Experimental): The individuals of the group received 5 treatments in total for 10 minutes that included: posterior to anterior spinal accessory mobilization passive physiological inter vertebral rotation The above was applied to the level that the MRI showed disc degeneration
  Interventions: Procedure: spinal mobilization
- Sham Treatment (Sham Comparator): The investigator touched the skin overlying the low back statically for 10 minutes
  Interventions: Procedure: sham treatment
- Classic Physiotherapy (Active Comparator): This group received static hamstring stretch for 5 minutes, TENS (2 channels biphasic pulse, 90Hz, 100μs pulse width) for 20 minutes and 15 minutes of Swedish type massage (effleurage, petrissage, kneading)
  Interventions: Device: TENS; Procedure: swedish type massage; Procedure: static hamstring stretch

INTERVENTIONS:
Device: TENS — Enraf-Nonius Sonopuls 692
  Arms: Classic Physiotherapy
Procedure: spinal mobilization — passive physiological intervertebral movements and passive accessory posteroanterior mobilization
  Arms: Spinal mobilization
Procedure: swedish type massage — petrissage, effleurage, tapotement
  Arms: Classic Physiotherapy
Procedure: static hamstring stretch — static hamstring stretching
  Arms: Classic Physiotherapy
Procedure: sham treatment — touching of the skin overlying the lumbar area
  Arms: Sham Treatment

SUMMARY:
Introduction: patients with chronic back pain as a result of degenerated disc disease, besides pain also present with impaired gait. The purpose of this study is to evaluate both the clinical data using clinical rating scales, such as Oswestry Disability Index Greek version (ODI), Numerical Pain Rating Scale for low back pain and leg pain (NPRS) and the Roland Morris Disability Questionnaire Greek Version, and kinetic and kinematic characteristics during gait analysis in patients with chronic low back pain as a result of the degenerated disc disease (Disc Degenerative Disease), before and after application of manual therapy techniques.

Methodology: for the purposes of the study, 75 patients suffering from chronic low back pain were randomly divided into 3 groups of 25 each. Each group received five sessions with the first group receiving manual therapy treatment (spinal mobilisation), the second a sham treatment and the third, classic physiotherapy (stretching exercises, TENS and massage). To evaluate the effectiveness of each treatment, the visual analog pain scale, two questionnaires (Oswestry and Roland Morris) and also an optoelectronic system for recording and analysis of gait (kinetic and kinematic data) were utilized.

DETAILED DESCRIPTION:
This was a randomized controlled trial comparing the efficacy of spinal mobilization with other physiotherapy interventions (stretching, TENS application and Swedish type massage) and sham treatment in a group of chronic low back pain patients. The outcome measures included three dimensional gait analysis (kinetic and kinematic data) as well as clinical indicators (numerical pain rating scale, Oswestry disability index, Roland-Moris Disability questionnaire).

ELIGIBILITY:
Inclusion Criteria:

* low back pain for over 3 months
* recent lumbar MRI (up to 12 months)
* able to walk without the need of walking aids

Exclusion Criteria:

* leg length discrepancy of over 2 cm
* history of spinal surgery
* history of autoimmune disease
* history of spondylolysis and spondylolisthesis
* spinal fractures
* pregnancy
* respiratory and/or cardiac disease
* history of stroke
* hip, knee or ankle osteoarthritis
* cauda equina syndrome
* spinal inflammation
* spinal tumor
* steroid drug use in the last month
* osteoporosis

Ages: 21 Years to 78 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2011-12; Primary Completion 2014-10 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GEORGIOS O KREKOUKIAS, PT, MSc, PhD, Principal Investigator — University of Ioannina; IOANNIS D GELALIS, MD, PhD, Study Director — University of Ioannina

IPD SHARING:
Plan to Share IPD: Yes
individual participant's grade of disc degeneration has been shared as an appendix in an already published article: http://dx.doi.org/10.1080/10669817.2016.1184435. Please note that no more IPD will be shared.

REFERENCES:
- [Background] Goodsell M, Lee M, Latimer J. Short-term effects of lumbar posteroanterior mobilization in individuals with low-back pain. J Manipulative Physiol Ther. 2000 Jun;23(5):332-42. PMID 10863253
- [Background] Managing chronic low back pain. How to avoid the problem, lower risk, and manage the discomfort when it occurs. Duke Med Health News. 2014 May;20(5):1-2. No abstract available. PMID 24960844
- [Background] Goel A, Loudon J, Nazare A, Rondinelli R, Hassanein K. Joint moments in minor limb length discrepancy: a pilot study. Am J Orthop (Belle Mead NJ). 1997 Dec;26(12):852-6. PMID 9413588
- [Background] Liu XC, Fabry G, Molenaers G, Lammens J, Moens P. Kinematic and kinetic asymmetry in patients with leg-length discrepancy. J Pediatr Orthop. 1998 Mar-Apr;18(2):187-9. PMID 9531400
- [Background] McCaw ST, Bates BT. Biomechanical implications of mild leg length inequality. Br J Sports Med. 1991 Mar;25(1):10-3. doi: 10.1136/bjsm.25.1.10. PMID 1913023
- [Background] Kawaguchi Y, Matsui H, Tsuji H. Back muscle injury after posterior lumbar spine surgery. Part 2: Histologic and histochemical analyses in humans. Spine (Phila Pa 1976). 1994 Nov 15;19(22):2598-602. doi: 10.1097/00007632-199411001-00018. PMID 7855687
- [Background] Taylor H, McGregor AH, Medhi-Zadeh S, Richards S, Kahn N, Zadeh JA, Hughes SP. The impact of self-retaining retractors on the paraspinal muscles during posterior spinal surgery. Spine (Phila Pa 1976). 2002 Dec 15;27(24):2758-62. doi: 10.1097/00007632-200212150-00004. PMID 12486343
- [Background] Wang D, Bergstrom E, Clarke M, Henderson N, Gardner B. Mobility of the spine after spinal surgery in acute spinal cord injury. Spinal Cord. 2003 Nov;41(11):593-9. doi: 10.1038/sj.sc.3101528. PMID 14569260
- [Background] O'Sullivan PB, Phyty GD, Twomey LT, Allison GT. Evaluation of specific stabilizing exercise in the treatment of chronic low back pain with radiologic diagnosis of spondylolysis or spondylolisthesis. Spine (Phila Pa 1976). 1997 Dec 15;22(24):2959-67. doi: 10.1097/00007632-199712150-00020. PMID 9431633
- [Background] Egerton T, Danoudis M, Huxham F, Iansek R. Central gait control mechanisms and the stride length - cadence relationship. Gait Posture. 2011 Jun;34(2):178-82. doi: 10.1016/j.gaitpost.2011.04.006. Epub 2011 May 7. PMID 21550245
- [Background] Mello RG, Oliveira LF, Nadal J. Digital Butterworth filter for subtracting noise from low magnitude surface electromyogram. Comput Methods Programs Biomed. 2007 Jul;87(1):28-35. doi: 10.1016/j.cmpb.2007.04.004. Epub 2007 Jun 4. PMID 17548125
- [Background] Love A, Leboeuf C, Crisp TC. Chiropractic chronic low back pain sufferers and self-report assessment methods. Part I. A reliability study of the Visual Analogue Scale, the Pain Drawing and the McGill Pain Questionnaire. J Manipulative Physiol Ther. 1989 Feb;12(1):21-5. PMID 2522493
- [Background] Moutzouri M, Billis E, Strimpakos N, Kottika P, Oldham JA. The effects of the Mulligan Sustained Natural Apophyseal Glide (SNAG) mobilisation in the lumbar flexion range of asymptomatic subjects as measured by the Zebris CMS20 3-D motion analysis system. BMC Musculoskelet Disord. 2008 Oct 1;9:131. doi: 10.1186/1471-2474-9-131. PMID 18828921
- [Background] Shrout PE, Fleiss JL. Intraclass correlations: uses in assessing rater reliability. Psychol Bull. 1979 Mar;86(2):420-8. doi: 10.1037//0033-2909.86.2.420. PMID 18839484
- [Background] Henriksen M, Lund H, Moe-Nilssen R, Bliddal H, Danneskiod-Samsoe B. Test-retest reliability of trunk accelerometric gait analysis. Gait Posture. 2004 Jun;19(3):288-97. doi: 10.1016/S0966-6362(03)00069-9. PMID 15125918
- [Background] Weir JP. Quantifying test-retest reliability using the intraclass correlation coefficient and the SEM. J Strength Cond Res. 2005 Feb;19(1):231-40. doi: 10.1519/15184.1. PMID 15705040
- [Result] Pivec R, Stokes M, Chitnis AS, Paulino CB, Harwin SF, Mont MA. Clinical and economic impact of TENS in patients with chronic low back pain: analysis of a nationwide database. Orthopedics. 2013 Dec;36(12):922-8. doi: 10.3928/01477447-20131120-04. PMID 24579210
- [Result] Shum GL, Tsung BY, Lee RY. The immediate effect of posteroanterior mobilization on reducing back pain and the stiffness of the lumbar spine. Arch Phys Med Rehabil. 2013 Apr;94(4):673-9. doi: 10.1016/j.apmr.2012.11.020. Epub 2012 Nov 23. PMID 23178541
- [Result] Bronfort G, Haas M, Evans R, Kawchuk G, Dagenais S. Evidence-informed management of chronic low back pain with spinal manipulation and mobilization. Spine J. 2008 Jan-Feb;8(1):213-25. doi: 10.1016/j.spinee.2007.10.023. PMID 18164469
- [Result] Kaufman KR, Miller LS, Sutherland DH. Gait asymmetry in patients with limb-length inequality. J Pediatr Orthop. 1996 Mar-Apr;16(2):144-50. doi: 10.1097/00004694-199603000-00002. PMID 8742274
- [Result] Thomas E, Silman AJ, Papageorgiou AC, Macfarlane GJ, Croft PR. Association between measures of spinal mobility and low back pain. An analysis of new attenders in primary care. Spine (Phila Pa 1976). 1998 Feb 1;23(3):343-7. doi: 10.1097/00007632-199802010-00011. PMID 9507623
- [Result] Callaghan JP, Patla AE, McGill SM. Low back three-dimensional joint forces, kinematics, and kinetics during walking. Clin Biomech (Bristol). 1999 Mar;14(3):203-16. doi: 10.1016/s0268-0033(98)00069-2. PMID 10619108
- [Result] Chao EY, Laughman RK, Schneider E, Stauffer RN. Normative data of knee joint motion and ground reaction forces in adult level walking. J Biomech. 1983;16(3):219-33. doi: 10.1016/0021-9290(83)90129-x. PMID 6863337

RESULTS

PARTICIPANT FLOW:
Groups:
- Classic Physiotherapy: This group received static hamstring stretch for 5 minutes, TENS (2 channels biphasic pulse, 90Hz, 100μs pulse width) for 20 minutes and 15 minutes of Swedish type massage (effleurage, petrissage, kneading)
  Transcutaneous electrical nerve stimulation: Enraf-Nonius Sonopuls 692
  swedish type massage: petrissage, effleurage, tapotement
  muscle stretching: static hamstring stretching
Period: Overall Study
Arm/Group | Spinal Mobilization | Sham Treatment | Classic Physiotherapy
Started | 25 | 25 | 25
Completed | 25 | 25 | 25
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Spinal Mobilization; Sham Treatment; Classic Physiotherapy: The individuals of the group were asked to fill-in the Roland-Morris and the Oswestry questionnaires. The researcher assessed the baseline pain using the numerical pain rating scale. In addition, the gait of all subjects was assessed using 3D kinematic analysis and force platforms to assess kinetic values.
- Total: Total of all reporting groups
Arm/Group | Spinal Mobilization | Sham Treatment | Classic Physiotherapy | Total
Number analyzed (Participants) | 25 | 25 | 25 | 75
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 20 | 22 | 19 | 61
  >=65 years | 5 | 3 | 6 | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.96 (16.07) | 50.08 (12.61) | 45.48 (14.58) | 47.5 (14.58)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 11 | 9 | 33
  Male | 12 | 14 | 16 | 42
Region of Enrollment [Number; unit: participants]
  Greece | 25 | 25 | 25 | 75

OUTCOME MEASURES:

1. Primary Outcome: Change in the Numerical Pain Rating Scale
Description: this scale expresses the self rated pain levels in a 0 to 10 range with 0 meaning no pain and 10 the worst imaginable pain.
Time Frame: before the beginning, after the end of 5 weeks and 6 months after the last treatment session for each patient
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Spinal Mobilization | Sham Treatment | Classic Physiotherapy
Number analyzed (Participants) | 25 | 25 | 25
units on a scale
  Baseline values | 5.96 (1.37) | 6.12 (1.05) | 6 (1)
  5 sessions after | 1.22 (1.1) | 5.88 (0.92) | 4.96 (0.89)
  6 months after | 1.32 (0.75) | 6.02 (0.93) | 5.08 (0.95)

2. Primary Outcome: Change in the Oswestry Low Back Pain Disability Index
Description: this is a self rated questionnaire that is expressed in a percentage with 0% meaning no disability and 100% meaning total disability. The minimum detectable change is reported to be 10% points
Time Frame: before the beginning, after the end of 5 weeks for each patient and 6 months after the last treatment session for each patient
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Spinal Mobilization | Sham Treatment | Classic Physiotherapy
Number analyzed (Participants) | 25 | 25 | 25
units on a scale
  Baseline values | 33.28 (15.02) | 32 (8.32) | 31.04 (11.07)
  5 sessions after | 9.84 (3.87) | 31.76 (8.51) | 27.28 (9.53)
  6 months after | 8.96 (3.75) | 32.8 (8.64) | 28.56 (9.62)

3. Primary Outcome: Change in the Roland-Morris Disability Questionnaire
Description: The Roland-Morris Disability Questionnaire is designed to assess self-rated physical disability caused by low back pain. The Roland-Morris Disability Questionnaire is most sensitive for patients with mild to moderate disability due to acute, sub-acute or chronic low back pain.
  For patients with severe disability the Oswestry disability questionnaire is recommended. in this case, we used the 24 question version in which 0 means no disability and 24 means total disability.
Time Frame: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Spinal Mobilization | Sham Treatment | Classic Physiotherapy
Number analyzed (Participants) | 25 | 25 | 25
units on a scale
  Baseline values | 8.56 (3.56) | 10 (1.96) | 9.96 (3.19)
  5 sessions after | 2.44 (1.76) | 10.04 (2.05) | 8.76 (2.96)
  6 months after | 2.48 (1.29) | 10.23 (1.89) | 8.68 (2.87)

4. Primary Outcome: Change in the 3 Dimensional Gait Characteristics (Kinetic and Kinematic) (Motion Analysis Optoelectronic Gait Analysis System Along With 2 Kistler Force Platforms)
Description: The data was recorded using relevant software (Cortex, Calcium Solver, Skeleton Builder, DV Reference, Sky Scripting, KinTools RT). Κinetic and kinematic data were assessed and analysed at 3 different gait cycle time moments defined by the gait cycle and the amount of ground reaction force (GRF) during both left and right foot contact: moment 1 (T1) was at maximum GRF during heel strike, moment 2 (T2) at minimum GRF during mid stance, and moment 3 (T3) at maximum GRF during acceleration before toe off (http://www.oandplibrary.org/popup.asp?frmItemId=2A1E740F-13FD-4A68-B8A3-83A407795B5F&frmType=image&frmId=1). From these, we extrapolated the quotient (between R and L kinetic and kinematic data) values. A value of 1 would mean absolute symmetry between left and right side (Seliktar and Mizrahi, 1986). the participants walked for 10 times and the mean values of the best 3 measurements were used for analysis.
Time Frame: before the beginning and after the end of 5 weeks for each patient
Population: all participants were chronic low back pain patients with a variable degree of vertebral disc degeneration defined by the modified Pfirrmann scale
Measure: Mean (Standard Deviation); unit: quotient: degrees/degrees=no unit
Arm/Group | Spinal Mobilization | Sham Treatment | Classic Physiotherapy
Number analyzed (Participants) | 25 | 25 | 25
quotient: degrees/degrees=no unit
  torso position frontal plane quotient at T1 | -1.147 (0.035) | 0.852 (0.25) | -0.4 (0.18)
  torso position frontal plane quotient at T2 | -1.307 (0.127) | 0.172 (0.025) | -0.429 (0.33)
  pelvis position frontal plane quotient at T2 | 0.844 (0.102) | 1.295 (0.355) | 1.044 (0.422)
  torso position coronal plane quotient at T2 | 0.272 (0.058) | 1.645 (0.454) | -1.819 (0.485)
  pelvis position frontal plane quotient at T3 | -1.236 (0.232) | -0.16 (0.128) | -0.679 (0.254)

ADVERSE EVENTS:
Arm/Group | Spinal Mobilization | Sham Treatment | Classic Physiotherapy
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 0/25 | 0/25 | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No